CLINICAL TRIAL: NCT04377009
Title: A Randomized, Controlled, Blinded Study of Internet-guided Cognitive Behavioral Therapy for Insomnia in Military Service Members With History of Traumatic Brain Injury
Brief Title: Internet-guided Cognitive Behavioral Therapy for Insomnia in Military Service Members With History of TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNRM-02-9662
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Insomnia Chronic; Mild Traumatic Brain Injury
Keywords: Cognitive Behavioral Therapy; Insomnia; Concussion; Mild Traumatic Brain Injury
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active CBT-I (Experimental): Internet-guided cognitive behavioral therapy
  Interventions: Device: Sleep Healthy Using the Internet (SHUTi)
- Control (Other): Education control program
  Interventions: Other: Education Control Program

INTERVENTIONS:
Device: Sleep Healthy Using the Internet (SHUTi) — Cognitive behavioral therapy delivered via internet-guided program customized for military service members
  Arms: Active CBT-I
Other: Education Control Program — Online portal designed to inform participants about healthy lifestyle activities and general insomnia information
  Arms: Control

SUMMARY:
This study aims to validate an established internet-guided cognitive behavioral therapy for insomnia (CBT-I) as an alternative program to traditional in-person therapy that may increase treatment availability and utilization within the military health system. The version of the internet-guided CBT-I program being studied has been customized specifically for military service members.

The study will assess if the customized internet-guided CBT-I program will positively improve clinical measures of insomnia and quality of life outcomes in active or retired service members with primary insomnia and associated mild traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) represents a major health problem in United States military service members. Mild traumatic brain injury, also called "concussion", accounts for approximately 90% of the overall cases of TBI. Mild TBI (mTBI) is associated with various debilitating symptoms, such as headache, mood disorders, and sleep alterations. A high percentage of service members and veterans with suspected or confirmed mTBI are also diagnosed with insomnia or other sleep disorders.

In-person cognitive behavioral therapy for insomnia (CBT-I) has been documented as an effective therapy for treating insomnia. However, implementation within the Military Healthcare System (MHS) has been lacking due to lack of appropriately trained practitioners. Additionally, patients may overlook in-person therapy due to significant time commitment.

This study is a double-blind, randomized, controlled clinical trial to assess internet-guided CBT-I in military service members with insomnia and mTBI. The primary outcome measure for efficacy is the Insomnia Severity Index (ISI) with secondary cross-validation using the Pittsburgh Sleep Quality Index (PSQI). Approximately 200 participants will be randomized to treatment or control groups. Participants receiving active CBT-I will follow a 9-week internet-guided program requiring daily follow-up through an online portal that may be accessed via computer or phone. Participants in the control group will also receive access to an online portal for 9 weeks.

Primary analysis is percent improvement in severity symptoms assessed pre- and post-treatment. Secondary analysis is percent retained improvement in severity of symptoms assessed post-treatment and long-term follow-up at 6 months.

Secondary outcome measures will capture a variety of known and suspected insomnia precursors, predictors, or correlates and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Service member or veteran
* Ability to provide electronic informed consent and follow study-related instructions
* Presence of clinical insomnia for a period of at least 1 month prior to consent as confirmed by self-reported Insomnia Severity Index (ISI) score ≥15 and Pittsburgh Sleep Quality Index ≥5
* History of mild traumatic brain injury ≥6 months prior to consent, including blast-related, as confirmed by a telephone administered traumatic brain injury screener
* Reliable access to a telephone and the Internet via their computer or smartphone
* Stable regimen of medications for sleep or potentially affecting sleep over prior 1 month as confirmed by clinical history review

Exclusion Criteria:

* Current or previous cognitive behavioral therapy for insomnia (CBT-I) or electronic CBT- I intervention; participants may still receive other approved therapies provided via standard of care
* Life expectancy of <6 months
* Rapidly progressive illnesses (i.e., late-stage cancer, neurodegenerative conditions, major organ failure, etc.)
* Self-reported history of moderate to severe substance use disorders with the exception of nicotine
* Active bipolar disorder or psychosis that could be worsened by mild sleep restriction as part of electronic CBT-I
* Routine irregular work schedules or sleep patterns defined as shift work greater than 1 day per week
* Any other considerations that in the view of the principal investigator may adversely affect patient safety, participation, or scientific validity of the data being collected

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline and 9 weeks
  Comparison of changes in ISI scores from baseline to post-intervention. A clinically meaningful change will be defined as >=25% reduction in total symptom score.
Insomnia Severity Index (ISI) | Baseline and 3 months
  Comparison of changes in ISI scores from baseline to post-intervention. A clinically meaningful change will be defined as >=25% reduction in total symptom score.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | Baseline and 9 weeks
  Comparison of changes in PHQ-9 scores from baseline to post-intervention
Patient Health Questionnaire 9 (PHQ-9) | Baseline and 3 months
  Comparison of changes in PHQ-9 scores from baseline to post-intervention
PTSD Checklist for DSM-5 (PCL-5) | Baseline and 9 weeks
  Comparison of changes in PCL-5 scores from baseline to post-intervention
PTSD Checklist for DSM-5 (PCL-5) | Baseline and 3 months
  Comparison of changes in PCL-5 scores from baseline to post-intervention
Migraine Disability Assessment (MIDAS) | Baseline and 9 weeks
  Comparison of changes in MIDAS scores from baseline to post-intervention
Migraine Disability Assessment (MIDAS) | Baseline and 3 months
  Comparison of changes in MIDAS scores from baseline to post-intervention
Pittsburgh Sleep Quality Index (PSQI) | Baseline and 9 weeks
  Comparison of changes in PSQI scores from baseline to post-intervention
Pittsburgh Sleep Quality Index (PSQI) | Baseline and 3 months
  Comparison of changes in PSQI scores from baseline to post-intervention
Pittsburgh Sleep Quality Index (PSQI) with Addendum for PTSD (PSQI-A) | Baseline and 9 weeks
  Comparison of changes in PSQI-A scores from baseline to post-intervention
Pittsburgh Sleep Quality Index (PSQI) with Addendum for PTSD (PSQI-A) | Baseline and 3 months
  Comparison of changes in PSQI-A scores from baseline to post-intervention
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Baseline and 9 weeks
  Comparison of changes in FACIT-F scores from baseline to post-intervention
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Baseline and 3 months
  Comparison of changes in FACIT-F scores from baseline to post-intervention

OTHER OUTCOMES:
Sleep outcomes | 9 weeks; 3 months
  Assess changes in sleep outcomes and calculated sleep efficiency: bed time, sleep onset latency, number of awakenings, total duration of awakenings, wake time, arising time, daytime naps, soundness of sleep, sleep quality, sleep medication and alcohol use
Blinding efficacy | 3 months
  Assess investigator blinding efficacy as reflected by mid-intervention and post-intervention questionnaires
Concurrent Medications | 9 weeks; 3 months
  Assess concurrent medications and correlation with intervention efficacy
Participant Expectations | Baseline; 9 weeks; 3 months
  Assess participant expectation of benefit and blinding efficacy as reflected by pre-intervention and post-intervention questionnaires
Participant satisfaction | 3 months
  Assess participant satisfaction and help-seeking behavior as reflected by a 3-month follow-up questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David L Brody, MD, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Uniformed Services University, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifier-free participant data sets will be shared with the Uniformed Services University Center for Neuroscience and Regenerative Medicine Data Repository. Identifier-free data sets may also be shared with the Federal Interagency Traumatic Brain Injury Research (FITBIR) Data Repository.
Time Frame: After study completion, data sets will be de-identified and shared with the repositories. De-identified data sets will be stored in the repositories indefinitely.
Access Criteria: Access to the CNRM Data Repository will be determined b the CNRM Data Quality, Access, and Publication Committee. Investigators requesting access to the data will provide a list of investigators and collaborators who will have access to the data, documentation of Ethical Conduct of Research and Human Participants Protection Training, and documentation of Institutional Review Board Approval of the research project.
  Access to FITBIR will follow FITBIR Access Criteria
URL: https://fitbir.nih.gov/content/access-data

REFERENCES:
- [Derived] Malarkey ME, Fu AJ, Mannan N, Shaw OM, Haight TJ, Cota MR, Jahed NC, Werner JK, Brody DL. Internet-Guided Cognitive Behavioral Therapy for Insomnia Among Patients With Traumatic Brain Injury: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2420090. doi: 10.1001/jamanetworkopen.2024.20090. PMID 38980675

DOCUMENTS (1):
  • Informed Consent Form (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT04377009/ICF_000.pdf